CLINICAL TRIAL: NCT07075627
Title: An Observational Study to Evaluate the Incidence of Clinically Suspicious Lambert-Eaton Myasthenic Syndrome (LEMS) in Subjects Diagnosed With Small Cell Lung Cancer (SCLC)
Brief Title: A Study to Evaluate the Incidence of Clinically Suspicious Lambert-Eaton Myasthenic Syndrome (LEMS) in Subjects Diagnosed With Small Cell Lung Cancer (SCLC)
Status: Not yet recruiting | Type: Observational
Sponsor: Addario Lung Cancer Medical Institute (Other)
Responsible Party: Sponsor
Other Study IDs: ALCMI-024
Record Dates: First submitted 2025-07-11; First posted 2025-07-20 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Small Cell Lung Cancer ( SCLC ); Lambert Eaton Myasthenic Syndrome (LEMS)
Keywords: SCLC; LEMS; small cell lung cancer; lambert eaton myasthenic syndrome
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lambert-Eaton Myasthenic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SCLC: Diagnosis of SCLC within 1 year of enrollment

SUMMARY:
This is a multi-center observational study in subjects with a diagnosis of small cell lung cancer. Screening and/or medical record review for symptoms associated with Lambert Eaton Myasthenic Syndrome (LEMS) will be conducted.

DETAILED DESCRIPTION:
This is a multi-center observational study in subjects with a diagnosis of small cell lung cancer. All eligible subjects enrolled will undergo a brief, symptom directed neurological evaluation and VGCC antibody testing (to be performed at a participating Quest laboratory). The results (positive/negative) of VGCC antibody testing will be documented as well as the receptor type P, Q or N.

These tests will be repeated quarterly (Q3 months) for the duration of the study.

If at any visit the subject is found to be BOTH neurologically suggestive of having LEMS and the VGCC Ab test is positive, then the subject is considered to be Clinically Suspicious of having LEMS. At any visit if a subject meets the criteria of Clinically Suspicious of LEMS. the end of study visit will be completed. Once the End of study visit is completed no further treatment information will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men or women meeting Age of Majority (AOM) at the time of consent
2. Provide voluntary consent to participate in this study, documented via a signed informed Consent Form (ICF)
3. Any diagnosis of SCLC
4. Willing to provide clinical and medical information related to his/her cancer diagnoses to the study team as required
5. Willing to comply with the requirements of the study

Exclusion Criteria:

1. Has been diagnosed with non-tumor Lamber-Eaton Myasthenic syndrome (LEMS) > 1 year prior to the SCLC diagnosis.
2. Known existence of an uncontrolled intercurrent illness including, but not limited to, psychiatric illness or social situations that would impair compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: United States
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Suspicious LEMS | 1 year
  Incidence of clinically suspicious LEMS diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Sands, MD, Principal Investigator — Dana-Farber Cancer Institute; Gilbert Youssef, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol (2025-06-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT07075627/Prot_000.pdf